CLINICAL TRIAL: NCT06708143
Title: Noninvasive Temporal Interference Stimulation for the Treatment of Drug Resistant Epilepsy
Brief Title: Temporal Interference for Drug Resistant Epilepsy
Acronym: TIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-316-002
Record Dates: First submitted 2024-11-23; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Drug Resistant Epilepsy
Keywords: Temporal Interference; Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal Interference (Experimental): The investigators perform temporal interference (TI) stimulation to patients with drug-resistant epilepsy. They observe clinical manifestations before, during, and after stimulation to investigate the efficiency of TI.
  Interventions: Other: Temporal Interference

INTERVENTIONS:
Other: Temporal Interference — Researchers apply temporal interference (TI) stimulation to the deep brain nuclei of drug resistant epilepsy patients.
  Other Names: TI

SUMMARY:
This single-center prospective study aims to investigate the treatment efficacy of temporal interference (TI) in drug-resistant epilepsy patients aged 6-60.

DETAILED DESCRIPTION:
Temporal Interference (TI) technology is a novel non-invasive method for deep brain stimulation (DBS). By generating an overlapping electric field from safe currents, TI creates focused stimulation in targeted deep brain areas. This approach allows for the exploration of deep brain nuclei functions and has the potential to serve as a non-invasive alternative to traditional invasive DBS for clinical treatments.

This study aims to investigate the treatment efficacy of TI deep brain stimulation by including drug-resistant patients aged 6-60. During and after TI stimulation, clinical and electrophysiology data will be recorded. Clinical, imaging and electrophysiology data will be analyzed and processed to advance the treatment of drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 6 -60 years of age.
* Patients must be clinically evaluated as having drug resistant epilepsy.
* Persistence of disabling seizures at least 2 times per months or greater.
* Informed consent signed.

Exclusion Criteria:

* Psychogenic non-epileptic seizures within 12 months;
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., pacemaker, spinal cord stimulator, responsive neurostimulation) or any metallic implants in the head (e.g., aneurysm clips, cochlear implants). Note: Vagal nerve stimulators are allowed if the parameter remains stable for at least 3 months prior to the screening visit;
* Risk factors that would put the participant at risk for intraoperative or postoperative bleeding. (e.g., coagulation abnormalities, etc.) or the need for chronic anticoagulation or antiplatelet aggregation medications; IQ < 55 or severe cognitive dysfunction, unable to complete the study; Diagnosed with a progressive neurological disorder (including progressive Rasmussen's encephalitis, etc.);
* Diagnosed with a severe neuropsychiatric disorder such as dementia, major depression (admission to a psychiatric specialty/hospital within 5 years or any suicidal or self-injurious tendencies), schizophrenia, or neurodegenerative disorders;
* Diagnosed with other serious physical disorders, internal diseases or severe abnormalities in liver or kidney function; Pregnant, or planning to pregnant within 2 years; Participation in another clinical study within 3 months; Not suitable for enrollment as assessed by the multidisciplinary team of the center.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency (SF28) | Up to 1 year after TI stimulation
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as mean of 3- month SF28 in the baseline period. The seizure frequency in double-blind phase is defined as SF28 per month during the double-blind period. Percent change in seizure frequency=100*(double-blind SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 1 year after TI stimulation
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Life quality evaluation | Up to 1 year after TI stimulation
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score. The minimum and maximum values, and whether higher scores mean a better or worse outcome.
Cognitive function evaluation (MMSE) | Up to 1 year after TI stimulation
  Percentage change from baseline in Mini-Mental State Examination (MMSE) score. The MMSE score ranges from 0 to 30, with higher scores representing better cognitive function and lower scores indicating greater cognitive impairment.
Cognitive function evaluation (MoCA) | Up to 1 year after TI stimulation
  Percentage change from baseline in Montreal Cognitive Assessment (MoCA) score. The MoCA score ranges from 0 to 30, with higher scores indicating better cognitive function and lower scores suggesting greater cognitive impairment.
Adverse Events | Up to 1 year after TI stimulation
  Rate of adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Up to 1 year after TI stimulation
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China